CLINICAL TRIAL: NCT00894998
Title: Randomized Clinical Trial of Sodium Heparin Effectiveness and Security in Patients Submitted to Heart Surgery Using Bypass
Brief Title: Efficacy and Safety of Sodium Heparin in Patients (Cristália)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEPSBCCV0109_CRI; Heparin Cristália (Version 8)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Surgery
Keywords: heparin cardiac surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heparin sodium 5.000 UI - Cristália
  Interventions: Biological: heparin sodium - Cristália
- 2 (Active Comparator): Heparin Sodium 5.000 USP - APP
  Interventions: Biological: Heparin sodium APP

INTERVENTIONS:
Biological: heparin sodium - Cristália — Heparin sodium 5000UI - Cristália
  Arms: 1
Biological: Heparin sodium APP — Heparin Sodium 5.000 USP - APP
  Arms: 2

SUMMARY:
The objective of this study is to verify, through a randomized, single-blind, multicentre, parallel and comparative study, the effectiveness of heparin sodium of porcine origin in patients undergoing heart surgery at that require the aid of cardiopulmonary bypass, through the control of hemostasis during and after surgery, based on the strengths of markers of coagulation TCA, TTPA, Anti-Xa, heparin bioavailable and loss of excessive blood (bleeding) at the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree with all aspects of the study and sign the FICT;
* Patients of both sexes;
* Patients aged above 18 years;
* Patients with cardiac surgery and requiring movement; AND
* Extracorporeal.

Exclusion Criteria:

* Patients with hematological disorders that compromise the surgical changes (eg myeloproliferative syndromes, anemia Hb <11.0 g / dL,
* Platelets < 150,000 mm3);
* Patients with disorders of hemostasis (INR> 1.40) (rTTPA> 1.40);
* Patients with renal dysfunction (creatinine> 1.50);
* Patients with deep hyperthermia;
* Liver disease (AST and ALT> 2 times that of the reference value);
* Patients with a history of allergy to heparin or protamine;
* Patients with history of heparin-induced thrombocytopenia;
* Tables infection (eg endocarditis, infection of immune human (HIV), hepatitis B and C, septicemia and pneumonia);
* Reoperations;
* Use of antiplatelet (clopidogrel and ticlopidine) for less than 7 days;
* Use of acetylsalicylic acid is less than 5 days;
* Use of low molecular weight heparin for less than 24 hours; OR
* Use of non-fractioned heparin for less than 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of TTPA, Anti-Xa and ACT | Pre - Operative (T0) Pre Heparinization (T1) Top of Extracorporeal (T2) Period Intraoperative (T3) Termination Extracorporeal (T4) Postoperative
Comparison of bleeding | Pre - Operative (T0) Pre Heparinization (T1) Top of Extracorporeal (T2) Period Intraoperative (T3) Termination Extracorporeal (T4) Postoperative

SECONDARY OUTCOMES:
Adverse reactions | Pre - Operative (T0) Pre Heparinization (T1) Top of Extracorporeal (T2) Period Intraoperative (T3) Termination Extracorporeal (T4) Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil